CLINICAL TRIAL: NCT01969669
Title: A Phase 1 Study to Assess the Effect of Ketoconazole on the Pharmacokinetics of ABT-199
Brief Title: A Study to Assess the Effect of Ketoconazole on the Metabolism of ABT-199
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: M13-364
Record Dates: First submitted 2013-10-22; First posted 2013-10-25 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2014-10

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: non-Hodgkin's lymphoma; GDC-0199; Safety; Relapsed; Refractory; ABT-199; Pharmacokinetics; Cancer
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Recurrence; Neoplasms | interventions — venetoclax; Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm A (ABT-199 and ketoconazole) (Experimental)
  Interventions: Drug: ABT-199; Drug: Ketoconazole

INTERVENTIONS:
Drug: ABT-199 — Subjects will be dosed with ABT-199, then dosed with ABT-199 in combination with ketoconazole
  Other Names: GDC-0199
Drug: Ketoconazole — Subjects will be dosed with ABT-199, then dosed with ABT-199 in combination with ketoconazole

SUMMARY:
This is an open-label multicenter, study to assess the pharmacokinetic interaction of ketoconazole with ABT-199 in up to 12 subjects with relapsed or refractory non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
This is a Phase 1 study designed to assess how the body processes the study drug ABT-199 when taken alone and in combination with ketoconazole and to assess the safety of ABT-199 in combination with ketoconazole. Subjects may enroll in a separate extension study to continue receiving ABT-199 after completion of this study.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have relapsed or refractory non-Hodgkin's lymphoma.
* Subject must have histologically documented diagnosis of non-Hodgkin's lymphoma as defined by a B-cell neoplasm in the World Health Organization (WHO) classification scheme except as noted in the exclusion criteria.
* Subject has an Eastern Cooperative Oncology Group (ECOG) performance score of 0 to 2.
* Subject must have adequate bone marrow (independent of growth factor support per local laboratory reference range), coagulation, renal and hepatic function:

  * Absolute Neutrophil Count (ANC) greater than or equal to 1000/µL (without growth factor support unless neutropenia is clearly due to underlying disease);
  * Platelets greater than or equal to 75,000/mm3 (unless thrombocytopenia is clearly due to disease-related immune thrombocytopenia or to underlying disease; entry platelet count must be independent of transfusion within 14 days of Screening);
  * Hemoglobin greater than or equal to 9.0 g/dL (unless anemia is clearly due to underlying disease; entry hemoglobin must be independent of transfusion within 14 days of Screening);
  * If cytopenias are present, no evidence of myelodysplastic syndrome or hypoplastic bone marrow;
  * Subject must have activated partial thromboplastin time (aPTT) and prothrombin time (PT) not to exceed 1.5 × the upper normal limit (ULN);
  * Calculated creatinine clearance greater than or equal to 50 mL/min using a 24-hour urine collection for creatinine clearance or per the Cockcroft-Gault equation;
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less than or equal to 3.0 × ULN of institution's normal range;
  * Bilirubin less than or equal to 1.5 × ULN. Subjects with Gilbert's Syndrome may have a bilirubin greater than 1.5 × ULN per discussion with the AbbVie medical monitor.

Exclusion Criteria:

* Subject has been diagnosed with Post-Transplant Lymphoproliferative Disease (PTLD), Burkitt's lymphoma, Burkitt-like lymphoma, lymphoblastic lymphoma/leukemia, chronic lymphocytic leukemia (CLL), small lymphocytic lymphoma (SLL), or mantle cell lymphoma (MCL).
* Subject is receiving combination anti-retroviral therapy for HIV (due to potential drug-drug interactions between anti-retroviral medications and ABT-199, as well as anticipated ABT-199 mechanism based lymphopenia that may potentially increase the risk of opportunistic infections).
* Subject has hypersensitivity to ketoconazole.
* Subject has a cardiovascular disability status of New York Heart Association Class greater than or equal to 2. Class 2 is defined as cardiac disease in which patients are comfortable at rest but ordinary physical activity results in fatigue, palpitations, dyspnea or anginal pain.
* Subject has a significant history of renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, cardiovascular, or hepatic disease within the past 6 months that in the opinion of the investigator would adversely affect his/her participating in this study.
* Subject has malabsorption syndrome or other condition which precludes enteral route of administration (e.g., prior surgical resection).
* Subject has undergone an allogeneic stem cell transplant.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-12; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Determination of maximum observed plasma concentration (Cmax), time to Cmax (peak time, Tmax), terminal phase elimination rate constant (beta), terminal phase elimination half-life (t1/2), & area under the plasma concentration-time curve (AUC) of ABT-199 | Measured pre-dose and up to 96 hours post-dose ABT-199
  Blood samples for pharmacokinetic (PK) analysis of ABT-199 will be collected at designated timepoints to assess the PK parameters for ABT-199 alone relative to ABT-199 with ketoconazole

SECONDARY OUTCOMES:
Number of subjects with adverse events | Measured up to 30 days after the last dose of study drug
  Subjects will be monitored for clinical and laboratory evidence of adverse events throughout the study
Percentage of subjects with adverse events | Measured up to 30 days after the last dose of study drug
  Subjects will be monitored for clinical and laboratory evidence of adverse events throughout the study
Change in physical exam finding, including vital signs | Measured from Day 1 up to 30 days after the last dose of study drug
  Body temperature, weight, blood pressure, heart rate
Change in clinical laboratory test results | Measured from Day 1 up to 30 days after the last dose of study drug
  Chemistry, coagulation, hematology, urinalysis
Change in cardiac assessment findings | Measured from Day 1 up to Day 12
  Electrocardiogram

CONTACTS AND LOCATIONS:
Overall Officials: David Chien, MD, Study Director — AbbVie
Locations (3):
- United States (3):
  - Site Reference ID/Investigator# 97498, Tucson, Arizona
  - Site Reference ID/Investigator# 92593, Lebanon, New Hampshire
  - Site Reference ID/Investigator# 101415, Hackensack, New Jersey

REFERENCES:
- [Result] Agarwal SK, Salem AH, Danilov AV, Hu B, Puvvada S, Gutierrez M, Chien D, Lewis LD, Wong SL. Effect of ketoconazole, a strong CYP3A inhibitor, on the pharmacokinetics of venetoclax, a BCL-2 inhibitor, in patients with non-Hodgkin lymphoma. Br J Clin Pharmacol. 2017 Apr;83(4):846-854. doi: 10.1111/bcp.13175. Epub 2017 Jan 18. PMID 27859472